CLINICAL TRIAL: NCT01880892
Title: Laryngopharyngeal Reflux Before and After Cricopharyngeal Myotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David G. Lott, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-010052
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Laryngopharyngeal Reflux; Zenker's Diverticulum
MeSH Terms: conditions — Laryngopharyngeal Reflux; Zenker Diverticulum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post cricopharyngeal myotomy (Experimental): Subjects scheduled to undergo an endoscopic criocopharyngeal myotomy, which is the standard treatment for a Zenker's diverticulum, will have levels of laryngopharyngeal reflux measured after the procedure.
  Interventions: Procedure: Cricopharyngeal myotomy; Diagnostic Test: PH probe Testing

INTERVENTIONS:
Procedure: Cricopharyngeal myotomy — Endoscopic laser cricopharyngeal myotomy is one of the standard treatments for Zenker's Diverticulum. It takes about 30 minutes and at our institution requires a one night of observation in the hospital.
Diagnostic Test: PH probe Testing — 24 hour PH probe testing, which will measure acid reflux following cricopharyngeal myotomy.

SUMMARY:
The purpose of this study is to see if people with reflux with a Zenker's diverticulum have increased reflux into the throat following a cricopharyngeal myotomy.

DETAILED DESCRIPTION:
Gastroesophageal reflux is considered to be a common cause of cricopharyngeal dysfunction and Zenker's diverticulum. In patients with severe symptoms of dysphagia, we perform a cricopharyngeal myotomy to release the tension at the upper esophageal sphincter. There has been some speculation that if the upper esophageal sphincter is severed, there could be an increase in reflux into the pharyngeal and laryngeal structures. The current gold standard for measuring laryngopharyngeal reflux (LPR) is 24 hour monitoring with a dual-electrode pH catheter. A newer device specifically measures LPR by sitting in the nasopharynx. The probe has been verified as accurate by several studies, with some postulating that since its recording intervals are closer together, it may be more accurate for measuring LPR. We aim to measure LPR with the new pH probe in patients with gastroesophageal reflux before and after cricopharyngeal myotomy to see if LPR becomes present or worsens after surgery.

All patients presenting with cricopharyngeal dysfunction or Zenker's diverticulum with a diagnosis or symptoms of gastroesophageal reflux or laryngopharyngeal reflux will be asked to participate in the study. If they meet the inclusion criteria, agree to participate, and wish to undergo surgery for their dysphagia, a baseline 24 hr laryngopharyngeal reflux study will be obtained using the Restech probe. Additionally, baseline dysphagia and reflux questionnaires will be obtained and an exam with flexible nasopharyngoscopy will be done. This exam is considered part of a standard exam for this condition and would be performed even if patients were not part of the research study. The surgical procedure will treat their dysphagia no differently than if they were not participating in the study. The patient will have their standard postoperative visit at 4 weeks, where their reflux and dysphagia symptoms will be assessed with questionnaires and a reflux finding score will be calculated via nasopharyngoscopy. At 3 months, an additional 24 laryngopharyngeal reflux study will be conducted with the Restech probe, and the patient will be seen in clinic for their final postoperative visit shortly thereafter. The questionnaires and the flexible nasopharyngoscopy for a reflux finding score will be repeated. The nasopharyngoscopy exam is standard of care for this patient visit. The patient would undergo the same number of nasopharyngoscopies even if they were not part of the study. During the study, if the patient is already on medication for reflux, they will be taken off their medication for 7 days in order to better detect changes in their LPR before and after cricopharyngeal myotomy. This is the standard protocol for patients being tested for LPR by the 24 hr pH probe study with the Restech probe. The patients will serve as their own controls as we are looking for significant increases in the amount of laryngopharyngeal reflux after cricopharyngeal myotomy. The data will be maintained in a database until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of gastroesophageal reflux
* presence of Zenker's diverticulum or cricopharyngeal hypertrophy
* undergoing surgery for Zenker's diverticulum or cricopharyngeal hypertrophy with endoscopic laser cricopharyngeal myotomy
* at least 18 years old

Exclusion Criteria:

* pregnant women
* children
* prisoners
* adults lacking capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Presence of LPR measured by: number of pH drops >3 standard deviations from baseline and the pharyngeal composite pH score. | 3 months postoperatively

SECONDARY OUTCOMES:
Reflux symptom index (RSI) score | 3 months postoperatively
Mayo Dysphagia Questionnaire Score | 3 months postoperatively
Reflux finding score | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: David Lott, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials